CLINICAL TRIAL: NCT03042182
Title: Open Label Trial of Therapeutic Vaccine in Patients With Cholangiocarcinoma
Brief Title: Trial of Therapeutic Vaccine in Patients With Cholangiocarcinoma
Acronym: cholangio
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immunitor LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03
Record Dates: First submitted 2017-01-26; First posted 2017-02-03 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2018-08

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Intervention Model Description: one arm open label study to last 2 months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single pill of V3-X vaccine administered once daily (Experimental): One pill of oral therapeutic vaccine V3-X administered to patients with cholangiocarcinoma for two months and changes in CA19.9 tumor marker from baseline levels versus post-treatment levels will be assessed as correlates of changes in tumor burden
  Interventions: Biological: Oral therapeutic vaccine V3-X to treat cholangiocarcinoma

INTERVENTIONS:
Biological: Oral therapeutic vaccine V3-X to treat cholangiocarcinoma — One single pill of V3-X vaccine administered once per day to patients with cholangiocarcinoma

SUMMARY:
Cholangiocarcinoma (CCA) is a malignant neoplasm originating from the epithelial cells lining the intra- or extrahepatic biliary ducts. It is the second-most common liver cancer, after hepatocellular carcinoma (HCC). About 6,000 people in the United States develop bile duct cancer each year. One-year survival is less than 25% and no effective and safe systemic treatments are currently available. Last year the completion of open-label phase 2 trial (NCT02256514) of hepcortespenlisimut-L (V5) has been reported, which has shown that two-third of Mongolian patients with advanced HCC had a favorable clinical response, including complete remissions and with overall survival over 90% after 1 year. So far a few patients with CCA were treated with V5, but it appeared that their response rate was somewhat inferior to patients with HCC since two (both with hemochromatosis) out six patients died within 6 months. In one patient who had improved clinically, the improvement was correlated with decrease in CA19-9 tumor marker, but no marker profile information is available in regard to other CCA patients. As V5 tablets are made from pooled blood of patients with HCC, in theory, they will be not very useful to patients with CCA. The goal of this project is to manufacture an immunotherapeutic formulation made from pooled heat- and chemically-inactivated blood from donors with CCA and initiate pilot open-label trial in 20 cholangiocarcinoma patients. This clinical trial will be conducted in collaboration with the National Cancer Center.

DETAILED DESCRIPTION:
Upon obtaining regulatory and ethical approvals the Phase II single-arm study will be initiated at the NCC involving 20 patients with confirmed CCA diagnosis. The trial will be short, it will last only 2 months, but this will be sufficient to gauge the safety and efficacy. Only those patients who have higher than normal levels of CA19-9 tumor marker will be enrolled, which will serve as a surrogate marker in a manner alpha fetoprotein (AFP) has been used as a predictor of clinical response in HCC patients. Additional primary endpoints will be overall survival and changes in tumor burden, with secondary endpoints being liver function tests and changes in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* only those positive for CA19.9

Exclusion Criteria:

* pregnant and lactating females

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2020-02-20 (Estimated); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
Changes in CA19.9 tumor marker induced by daily dose of oral vaccine V3-X of cholangiocarcinoma | 2 months
  open label trial of once daily tablet of V3-X vaccine

SECONDARY OUTCOMES:
safety of vaccine | 2 months
  toxicity or adverse side effects, such as diarrhea and vomiting, we would have graded them according to accepted standards, e.g., NCI CTEP CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: aldar bourinbaiar, MD/PhD, Study Director — Immunitor LLC
Locations (2):
- Mongolia (2):
  - Immunitor LLC, Ulaanbaatar, CA
  - National Cancer Center, Ulaanbaatar

IPD SHARING:
Plan to Share IPD: No